CLINICAL TRIAL: NCT06059118
Title: Repeat Difluoromethylornithine and High Dose Testosterone With Enzalutamide in Asymptomatic Patients With Metastatic Castration-Resistant Prostate Cancer: The APEX (Androgen and Polyamine Elimination Alternating With Xtandi) Trial
Brief Title: Difluoromethylornithine and High Dose Testosterone With Enzalutamide in Metastatic Castration-Resistant Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Panbela Therapeutics (Industry); Prostate Cancer Foundation (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J2326; IRB00371517 (Other: JHM IRB)
Record Dates: First submitted 2023-09-15; First posted 2023-09-28 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; metastatic prostate cancer; DFMO; Enzalutamide; High dose testosterone
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Eflornithine; testosterone 17 beta-cypionate; Gonadotropin-Releasing Hormone; Goserelin; Triptorelin Pamoate; luprolide acetate gel depot; Leuprolide; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; relugolix; enzalutamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Repeat Sequential DFMO and High dose Testosterone in Sequence with Enzalutamide (Experimental): Eligible patients will receive 7 days of DFMO (1000 mg PO bid) (days 1-7 of cycle), followed by 56 days of combined testosterone (testosterone cypionate 400 mg IM on day 8 and day 36) and DFMO (1000 mg PO bid) (days 8-63 of cycle), followed by 56 days of enzalutamide (160 mg PO daily) (days 64-119).
  Interventions: Drug: DFMO; Drug: testosterone cypionate; Drug: Luteinizing hormone-releasing hormone (LHRH) analogue; Drug: Enzalutamide

INTERVENTIONS:
Drug: DFMO — Each 119 day cycle, Days 1-7 patient will take 1000 mg by mouth (PO) twice a day (bid), and then on Day 8 - 63 patient will take 1000 mg PO bid while receiving high dose testosterone IM on Day 8 and Day 36 of cycle.
  Other Names: eflornithine; difluoromethylornithine
Drug: testosterone cypionate — On Day 8 and Day 36 of each 119 day cycle, patient will receive high dose testosterone at 400 mg through intramuscular (IM) injection.
  Other Names: DEPO-Testosterone Injection
Drug: Luteinizing hormone-releasing hormone (LHRH) analogue — Patients who have progressive disease after treatment with Abiraterone (Abi) will continue with androgen depravation therapy (ADT) with LHRH analogue (LHRH agonist drug (i.e. Zoladex, Trelstar, Eligard or Lupron) or LHRH antagonist drug (Degarelix or Relugolix)). Dosing instructions will vary between the different LHRH analogues. Patients should follow the dosing instructions as directed by their physician.
  Other Names: Zoladex; Trelstar; Eligard; Lupron; Degarelix; Relugolix
Drug: Enzalutamide — Each 119 day cycle, Days 64-119 patient will take 160 mg by mouth (PO) once a day (qd).
  Other Names: Xtandi

SUMMARY:
Asymptomatic patients with metastatic castrate resistant prostate cancer (mCRPC) without pain due to prostate cancer will be treated on an open label study to evaluate effectiveness of sequential treatment with the combination of difluoromethylornithine (DFMO) and high dose testosterone in sequence with enzalutamide to improve primary and secondary outcomes.

DETAILED DESCRIPTION:
Eligible patients are those with mCRPC who have progressive disease after treatment with Abiraterone (Abi) used as treatment for castration-sensitive or castration-resistant disease. Patients will continue on androgen deprivation therapy (ADT) with luteinizing hormone-releasing hormone (LHRH) agonist (i.e. Zoladex, Trelstar, Eligard, or Lupron) or LHRH antagonist (Degarelix or Relugolix) if not surgically castrated throughout the duration of the study to inhibit endogenous testosterone production. One cycle of treatment will be 119 days and will involve:

1. 7 days of DFMO at a dose of 1000 mg PO BID (D1-D7), followed by
2. 56 days of combined testosterone and DFMO (testosterone cypionate 400 mg IM on D8 and D36 with continued DFMO 1000 mg PO BID) (D8-D63), followed by
3. 56 days of enzalutamide (enzalutamide 160 mg PO daily) (D64-D119)

Patients will receive repeat cycles of treatment until clinical or radiographic progression or toxicity requiring drug cessation.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) Performance status ≤2.
2. Age ≥18 years.
3. Histologically-confirmed adenocarcinoma of the prostate.
4. Treated with continuous androgen ablative therapy (either surgical castration or LHRH agonist/antagonist).
5. Documented castrate level of serum testosterone (<50 ng/dl).
6. Metastatic disease radiographically documented by CT or bone scan.
7. Must have had disease progression while on abiraterone acetate based on:

   * PSA progression defined as an increase in PSA, as determined by 2 separate measurements taken at least 1 week apart And/ Or
   * Radiographic disease progression, based on RECIST 1.1 in patients with measurable soft tissue lesions or Prostate Cancer Working Group 3 (PCWG3) for patients with bone disease
8. Screening PSA must be ≥ 1.0 ng/mL.
9. Patients with soft tissue lesion amenable to biopsy must agree to biopsy collection pre-treatment and at a defined point on treatment to perform tumor tissue analysis.
10. Prior treatment with Provenge vaccine, 223Radium (Xofigo), Poly (ADP-ribose) polymerase (PARP) inhibitors, taxane chemotherapy, Lutetium prostate-specific membrane antigen (LuPSMA), antiandrogens (including enzalutamide, darolutamide, and apalutamide), and radiation is allowed if >4 weeks from last dose.
11. Prior treatment with bipolar androgen therapy (BAT) is allowed if the patient has progressed on an AR-axis inhibitor (i.e. abiraterone or antiandrogen) since BAT treatment.
12. Patients must be withdrawn from abiraterone for ≥ 2 weeks.
13. Attempts must be made to wean patients off prednisone prior to starting therapy. Patients who cannot be weaned due to symptoms may continue on lowest dose of prednisone achieved during weaning period.
14. Acceptable liver function:

    1. Bilirubin < 2.5 times institutional upper limit of normal (ULN)
    2. Aspartate transaminase (AST) (SGOT) and alanine transaminase (AST) (SGPT) < 2.5 times ULN
15. Acceptable renal function:

    Glomerular filtration rate (GFR) of 50 mL/min/1.73 m2 or higher. GFR will be estimated by the 2021 chronic kidney disease epidemiology (CKD-EPI) creatinine equation (REF: Inker LA, Eneanya ND, Coresh J, et al. Chronic Kidney Disease Epidemiology Collaboration. New Creatinine- and Cystatin C-Based Equations to Estimate GFR without Race. N Engl J Med 2021; 385:1737) using the online calculator found on UpToDate (https://www.uptodate.com/contents/calculator-glomerular-filtration-rate-gfr-by-ckd-epiequation-in-adults-conventional-and-si-units search=gfr&topicRef=2359&source=see_link).
16. Acceptable hematologic status:

    1. Absolute neutrophil count (ANC) ≥ 1500 cells/mm3 (1.5 ×109/L)
    2. Platelet count ≥ 100,000 platelet/mm3 (100 ×109/L)
    3. Hemoglobin ≥ 8 g/dL.
17. Ability to understand and willingness to sign a written informed consent document.
18. Sexually active participants with female partners of childbearing potential are eligible to participate if they agree to follow 1 of the following methods of contraception consistently, starting from screening, during the study and for at least 3 months after the last dose of DFMO and/or enzalutamide:

    * Are abstinent from penile-vaginal intercourse as their usual and preferred lifestyle (abstinent on a longterm and persistent basis) and agree to remain abstinent.
    * Are sterilized (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate);
    * Agree to use a male condom and have their partner use a contraceptive method with a failure rate of <1% per year as described below when having penile-vaginal intercourse with a woman of childbearing potential who is not currently pregnant, and who agrees to the use of a condom by her partner.

    In addition, participants must refrain from donating sperm starting from Screening, during the study and for at least 3 months after the last dose of DFMO and/or enzalutamide.
19. Sexually active participants with a pregnant or breastfeeding partner must agree to remain abstinent from penile-vaginal intercourse; or use a male condom during each episode of penile penetration during the study
20. Patients with soft-tissue disease amenable to biopsy as determined by Interventional Radiology must agree to serial biopsies as per the study schedule to be eligible.

Exclusion Criteria:

1. Pain due to metastatic prostate cancer requiring treatment intervention with opioid pain medication.
2. ECOG Performance status ≥3
3. Requirement for urinary self-catheterization for voiding due to obstruction secondary to prostatic enlargement well documented to be due to prostate cancer or benign prostatic hyperplasia (BPH).

   Patients with indwelling Foley or suprapubic catheter for obstructive symptoms are eligible.
4. Evidence of disease in sites or extent that, in the opinion of the investigator, would put the patient at risk from therapy with testosterone (e.g. femoral metastases with concern over fracture risk, severe and extensive spinal metastases with concern for spinal cord compression, extensive liver metastases).
5. Active uncontrolled infection. Patients with a history of HIV/AIDS may be eligible if CD4+ T cell (a type of lymphocyte that helps coordinate the immune response against infection and disease) counts are ≥ 350 cell/ul, they have had no opportunistic infection within the past 12 months, they have been on established antiretroviral therapy (ART) for at least four weeks, the HIV viral load is less than 400 copies/ml prior to enrollment, and there is no significant drug-drug interaction with ART and the study drugs. Patients with chronic hepatitis B (HBV) infection with active disease who meet criteria for anti HBV therapy are eligible if they are on a suppressive antiviral therapy prior to enrollment and there is no drug-drug interaction with the study drugs. Patients with a history of hepatitis C (HCV) infection are eligible if they have completed curative antiviral treatment and the HCV viral load is below the limit of quantification.
6. Any condition or mental impairment that may compromise the ability to give informed consent, patient's safety or compliance with study requirements as determined by the investigator.
7. Patients receiving anticoagulation therapy with warfarin, rivaroxaban, or apixaban are not eligible for study. [Patients on enoxaparin are eligible for study. Patients on warfarin, rivaroxaban, or apixaban, who can be transitioned to enoxaparin prior to starting study treatments will be eligible].
8. Patients are excluded with prior history of a thromboembolic event within the last 12 months that are not being treated with systemic anticoagulation.
9. Hematocrit >51%, untreated severe obstructive sleep apnea, uncontrolled or poorly controlled heart failure [per Endocrine Society Clinical Practice Guidelines (34)]
10. Patients allergic to sesame seed oil or cottonseed oil are excluded.
11. Major surgery (i.e., requiring general anesthesia) within 3 weeks before screening, or has not fully recovered from prior surgery (i.e., unhealed wound). Note: subjects with planned surgical procedures to be conducted under local anesthesia may participate.
12. Subjects with significant hearing loss defined as hearing loss that affects everyday life and/or for which a hearing aid is required.
13. Patients with history of seizure or any condition that may predispose to seizure (e.g., prior cortical stroke or significant brain trauma, brain arteriovenous malformation)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-04 (Actual); Primary Completion 2027-01-04 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
PSA response rate at Cycle 1 Day 64 | Cycle 1 Day 64 (each cycle is 119 days)
  Number of participants with >50% PSA decline from baseline by Cycle 1 Day 64.

SECONDARY OUTCOMES:
Progression-free survival | 3 years after end of treatment
  Time to radiographic or clinical progression or death.
PSA response rate at any timepoint | up to 13 months
  Number of participants with >50% PSA decline from baseline at any point on trial.
Safety as assessed by number of participants experiencing adverse events grade 3 or higher and serious adverse events. | 13 months
  Number of participants who experience adverse events grade 3 or high and serious adverse events, as defined by Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
PSA progression-free survival (PSA-PFS) | up to 13 months
  Time from the date of first dose to the time of PSA progression.
Measurable disease response rate | 13 months
  Number of participants with measurable disease with complete response or partial response per RECIST 1.1.
Pain Score | Up to 12 months
  The modified Patient-Reported Outcomes Measurement Information System (PROMIS) short form (SF) (v1.0 short forms 3a and 6b) pain scale is a validated self-reported instrument assessing average pain intensity and interference over the past 7-day period. Possible scores for each pain intensity questions range from 1 (no pain) to 5 (very severe) with higher scores reflecting higher pain intensity. Possible scores for each pain interference range from 1 (not at all) to 5 (very much) with higher scores reflecting higher pain interference.
Pain Score Change | Baseline, Up to 12 months
  Number of participants with changes in pain scores between baseline and post-treatment. Positive change scores are indicative of improvement in pain.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Sena, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University: Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No